CLINICAL TRIAL: NCT00463255
Title: Phase IV Interventional Study: Effect of Diet on Brain Function in Elderly Healthy People
Brief Title: Diet and the Aging Brain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ernaehrung-Neuromod 01
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Diet; elderly; age-related diseases; prevention; cognitive decline; Clinical study
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: diet

SUMMARY:
We investigate whether a change in diet could provide positive effects on general brain functions in healthy elderly people.

DETAILED DESCRIPTION:
The age-related degradation of cognitive functions even to the point of neurodegenerative disorders such as alzheimer's disease are a growing public-health concern with potentially devastating effects.

Refering to animal data and empirical studies, a healthy diet rich in unsaturated fatty acids and low in calories should improve cognitive functions such as learning and memory. To test this hypothesis, we study general brain functions in healthy elderly subjects (50-80 years old) during a short term diet.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* 50-80 years old
* moderate to heavy weight
* must be able to change diet at home

Exclusion Criteria:

* diabetes
* younger than 50 years
* BMI < 23
* already participating in other studys
* MMSE > 26
* eating disorders

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-08; Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
implicit visual-motor learning of a finger sequence of the hand.

SECONDARY OUTCOMES:
implicit learning of an artificial language
several plasma levels related to cognitive functions

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Knecht, MD, Prof., Study Chair — University Hospital Muenster; Bernd E Ringelstein, MD, Prof, Study Chair — University Hopsital Muenster; Agnes Floeel, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Department of Neurology, Münster, North Rhine-Westphalia, Germany